CLINICAL TRIAL: NCT04804722
Title: Risk of Developing Dementia and Associated Factors in Patients With Normal Brain FDG PET
Acronym: NOBET
Status: Completed | Type: Observational
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Principal Investigator, Antoine VERGER, MD, PhD, Central Hospital, Nancy, France
Other Study IDs: 2021PI044
Record Dates: First submitted 2021-03-16; First posted 2021-03-18 (Actual); Last update posted 2023-07-06 (Actual); Status verified 2023-07

CONDITIONS: Neurodegenerative Diseases; Cognitive Disorder
MeSH Terms: conditions — Neurodegenerative Diseases; Cognitive Dysfunction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: 18F-FDG PET-CT (fluorodesoxyglucose positron emission tomography) — 18F-FDG PET-CT exams during 30 minutes with injection of radiopharmaceutical product

SUMMARY:
Brain 18F-FDG PET (positron emission tomography) is recognised as having a good negative predictive value in the search for a neurodegenerative origin of cognitive disorders. Indeed, a ratio of 0.1 on the occurrence of worsening cognitive disorders has been reported in case of normal brain FDG PET.

However, the risk of developing objective cognitive disorders in patients with no cognitive complaints is estimated at 8% per year and the risk of developing dementia in patients with mild cognitive disorders at 22% per year.

Cerebral 18F-FDG PET is a prognostic factor for the occurrence of unusual clinical manifestations (MCI) or the conversion of MCI to Alzheimer's disease, but we do not really know the impact on the longer term occurrence of cognitive impairment in patients with normal cerebral 18F-FDG PET.

Only a longitudinal study will allow us to really know the true negative predictive value of a normal 18F-FDG PET scan and the factors associated with a risk of dementia in these subjects. This will allow us to better understand the prognostic impact of a normal brain 18F-FDG PET scan and to identify a sub-population that remains at risk, including in the case of normal brain 18F-FDG PET.

DETAILED DESCRIPTION:
Brain 18F-FDG PET is known to have a good negative predictive value in the search for a neurodegenerative origin to cognitive disorders. Indeed, a ratio of 0.1 on the occurrence of worsening cognitive disorders has been reported in case of normal brain FDG PET.

However, in patients without cognitive complaints, the risk of developing objective cognitive impairment is estimated to be 8% per year and the risk of developing dementia in patients with mild cognitive impairment 22% per year.

Brain 18F-FDG PET is a prognostic factor for the occurrence of MCI or for the conversion of MCI to Alzheimer's disease , but we do not really know the impact on the longer-term occurrence of cognitive impairment in patients with a normal brain 18F-FDG PET.

Also, it is commonly accepted that a normal brain 18F-FDG PET scan can rule out a neurodegenerative origin for cognitive impairment.

However, the detection sensitivity of brain 18F-FDG PET is about 90% . Furthermore, we do not know the pathophysiological factors that cause false negative PET scans and it would be interesting to study them (age, sex, medical history, results of neuropsychological tests, etc.).

Based on subjects available freely on the internet, an American team showed that brain 18F-FDG PET was predictive of cognitive decline in subjects with no or minor cognitive disorders.

Only a longitudinal study will allow to really know the true negative predictive value of a normal 18F-FDG PET scan and the factors associated with a risk of dementia in these subjects. This will allow us to better understand the prognostic impact of a normal brain 18F-FDG PET scan and to identify a subpopulation that remains at risk, including in case of normal brain 18F-FDG PET.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient who had a PET scan with 18F-FDG in the brain at least 3 years previously
* Patients referred for PET scans for cognitive disorders, whether or not they have been diagnosed
* Patients referred for PET scans for neurodegenerative pathology 18F-FDG PET brain scan interpreted as normal

Exclusion Criteria:

* Brain 18F-FDG PET scan considered abnormal after semi-quantitative analysis

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patient who had a PET scan with 18F-FDG in the brain at least 3 years previously for cognitive disorders or neurodegenrative pathology
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2022-01-20 (Actual); Primary Completion 2023-07-01 (Actual); Study Completion 2023-07-01 (Actual)

PRIMARY OUTCOMES:
Normal brain 18F-FDG PET | 3 years
  Number of patients with normal brain 18F-FDG PET who developed dementia with a clinical follow-up of at least 3 years

SECONDARY OUTCOMES:
Predictive parameters for the occurrence of dementia | 3 years
  Predictive parameters for the occurrence of dementia in patients with normal brain 18F-FDG PET with a clinical follow-up of at least 3 years

CONTACTS AND LOCATIONS:
Locations (1):
- Nuclear medicine Department CHRU de NANCY, Vandœuvre-lès-Nancy, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Heyer S, Simon M, Doyen M, Mortada A, Roch V, Jeanbert E, Thilly N, Malaplate C, Kearney-Schwartz A, Jonveaux T, Bannay A, Verger A. 18F-FDG PET can effectively rule out conversion to dementia and the presence of CSF biomarker of neurodegeneration: a real-world data analysis. Alzheimers Res Ther. 2024 Aug 13;16(1):182. doi: 10.1186/s13195-024-01535-3. PMID 39135067